CLINICAL TRIAL: NCT03675607
Title: Knowledge and Habitual Practices in the Preparation of Complementary Feeding in Spain a: Cross-sectional Study
Brief Title: Preparation of Complementary Feeding in Spain: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Academia Española de Nutrición y Dietética (Other)
Collaborators: LIDL España (Unknown)
Responsible Party: Sponsor
Other Study IDs: LIDL-PPIC-2018
Record Dates: First submitted 2018-06-11; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-06

CONDITIONS: Infant Nutritional Physiological Phenomena; Complementary Feeding
Keywords: Infant Nutritional Physiological Phenomena; Complementary feeding; Feeding Behavior; Food Preferences; Parenting; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Feeding Behavior; Food Preferences; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers infants <2years old: Caregivers of infants under 2 years of age (parents or other), of any gender, who prepare complementary feeding regularly (more than once a week).
  Interventions: Other: Complementary feeding behaviours

INTERVENTIONS:
Other: Complementary feeding behaviours — Any kind of complementary feeding practice
  Other Names: beikost use; baby-led weaning

SUMMARY:
Study design: Cross-sectional study, survey based

Study population: spanish people, caregivers of infants under 2 years old. Sample size: 1925 surveys.

Study duration and research process: 10 days on-line survey that will be opened through a launching page. The survey is composed of 3 blocks.

Statistical analysis: data will be analyzed using the Statistical Analysis System (SAS) package version 9.4 (or higher). The categorical variables will be presented in the form of lists of frequencies and percentages. For the quantitative variables (continuous or ordinal), indices of central tendency (mean, median) and dispersion (standard deviation and maximum and minimum values) will also be presented.

DETAILED DESCRIPTION:
Study design: cross-sectional study, survey to collect data about knowledge, opinions, attitudes or behaviors of the Spanish population in relation to the preparation of complementary feeding for children.

Study population: self-reported information will be collected from a sample of Spanish population. The participants will be people included in a Spanish private database (Netquest Iberia, more than 100,000 available panelists). This database is constituted as a closed panel, from which the participants are invited individually to carry out a survey, and are selected according to their characteristics and ideal representativeness for the purpose of the evaluation. The panel of participants has the International Organization for Standardization (ISO) 26362 certification, which represents the level of quality contrasted in methods of recruitment, and treatment of the panelist and the data. To reach the objective of this study, the calculation of the minimum representative sample of the Spanish population corresponds to the completion of 385 surveys in the national territory. However, in order to broaden the geographical diversity of the participants, and based on the characteristics of the panel used, the objective is to reach the maximum number of possible surveys in the observation period of the appropriate panelists (1,925 surveys in 10 days).

Duration of the study: the study begins once the on-line survey is made available to the participants. The survey is expected to be available for a period of 10 days.

Subsequently, the corresponding database will be closed and the results will be exploited. The total duration of the study, until the publication of objective results, is established in 6 months.

Research process: For the realization of this on-line survey, a closed database of 100,000 panelists will be used, from which the ideal profile of the participants will be selected and a personalized invitation will be issued for their participation.

Once the invitation to the candidates to participate has been issued, a period of availability of the 10-day on-line survey will be opened through a web portal. Each participant will enter said portal individually, through a unique, personalized and anonymous access code. Once the survey has been activated for a specific participant, and after a brief introductory information, the sociodemographic data will be requested to be tabulated in order to tabulate the overall results of the survey (Annex 1: BLOCK 1). After the completion of BLOCK 1, all participants will start BLOCK 2, in which, for those participants who indicate that they prepare complementary food based on "mainly shredded", they will be asked a discriminatory question (Do you prepare or have you elaborated porridges? If you answer negatively to this question, the participant will be directed to the information collection block (BLOCK 3), since it is not pertinent to assess their practice and opinion. However, the fact of having children or their age is not considered discriminatory for the completion of the entire survey, given that the opinion and methodology of people who by profession can prepare homemade porridges, even without children, (eg nursery workers), as well as the opinion of those who currently have no small children (eg over 50 years old) ), remains of interest for the main objective of the study. The data or sections corresponding to BLOCK 2 and BLOCK 3 are presented in Annexes 2 and 3, respectively. Participants can complete the survey sequentially, even from different terminals, always with the same access code. Once all the corresponding sections have been completed, the participant will validate the answers and confirm their final submission, at which time the data will be compiled in the global database corresponding to the collection of the information of all the completed surveys. At the end of the period of completing forms, the database will be closed and statistics will be exploited in order to obtain objective results.

Statistical analysis: the data will be analyzed using the statistical package SAS System version 9.4 (or higher). A descriptive statistic of all the variables collected will be made by completing the data collection form. The categorical variables will be presented in the form of lists of frequencies and percentages. For the quantitative variables (continuous or ordinal), indices of central tendency (mean, median) and dispersion (standard deviation and maximum and minimum values) will also be presented.

ELIGIBILITY:
Inclusion Criteria:

* people included in a Spanish private database (Netquest Iberia
* caregivers of infants <2years old who prepare at least complementary feeding twice a week (actual or in the past)
* any texture/type of complementary feeding (blended/beikost/solid)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Spanish people included in a Spanish private database (Netquest Iberia, more than 100,000 available panelists), constituted as a closed panel of caregivers of infants <2years old who prepare at least complementary feeding twice a week (actual or in the past). The panel of participants has the ISO 26362 certification, which represents the level of quality contrasted in methods of recruitment, panelization, treatment of the panelist and the data. In order to broaden the geographical diversity of the participants, and based on the characteristics of the panel used, the objective is to reach the maximum number of possible surveys in the observation period of the appropriate panelists (1,925 surveys in 10 days).
Sampling Method: Non-Probability Sample
Enrollment: 1925 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Texture/type of complementary feeding (dichotomic) | 1 month
  Know how caregivers prepare the complementary feeding, mainly blended or solid
Ingredient selection (%) | 1 month
  know how caregivers select ingredients to allow diversity
Food/ingredient amount (gr/100gr) | 1 month
  know the amount of food and ingredients are often used by caregivers
Ingredient preparation and cooking technique | 1 month
  know the ingredient preparation and cooking technique usually used by careguivers

SECONDARY OUTCOMES:
conservation technique | 1 month
  know what conservation techniques are used by caregivers
hygiene | 1 month
  mainly hand/ingrediente washing behaviours
Wold Health Organization (WHO) core indicators about complementary feeding | 1 month
  Wold Health Organization (WHO) core indicators about complementary feeding

CONTACTS AND LOCATIONS:
Locations (1):
- Academia Española de Nutrición y Dietética, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: within 6 months study completion